CLINICAL TRIAL: NCT03952793
Title: Development of the Organoids Technique From Metastases From Patients With Advanced Form of Prostate Cancer: Use in Basic Research
Brief Title: Organoids From Metastases of Prostate Cancer
Acronym: OrMePro
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility issues
Sponsor: Centre Antoine Lacassagne (Other)
Collaborators: Centre Méditerranéen de Médecine Moléculaire UMR_S-1065 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018/63
Record Dates: First submitted 2019-05-10; First posted 2019-05-16 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Extended biopsy
  Interventions: Other: extended biopsy

INTERVENTIONS:
Other: extended biopsy — Additional sample are performed during a biopsy to provide tumor tissues for the organoid technique development

SUMMARY:
The aim of the study is the development of the organoid culture technique from metastases from patients with advanced form of prostate cancer. Once the technique is set up, the organoid will serve to test several antitumor molecules.

ELIGIBILITY:
Inclusion Criteria:

* Patient with metastatic prostate cancer
* Patient having a biopsy programmed as part of his care.
* Patient having a biopsy programmed as part of hiscare.
* Patient with sufficient tumor volume after imaging data review by the radiologist to guarantee a sufficient quantity of material for the diagnosis of biopsy and additional material for the study.
* INR <1.5; Platelets > 50000 / μL

Exclusion Criteria:

* Patient under age of 18 years.
* Patient under Plavix or Effient or Ticlid without possibility of suspension for 5 days, low molecular weight heparin without possibility of suspension of the dose before the intervention, or Fondaparinux without possibility of suspension, or ReoPro without possibility of suspension for 24h and aPTT <50s and ACT <150s, or Integrilin or Aggrastat or Argatroban without possibility of suspension 4 H before the intervention, or Angiomax without possibility of suspending 2H to 3H if CrCL> 50 mL / min or 3H to 5h if CrCL <50 mL / min before the intervention or and Pradaxa without possibility of suspension 2 to 3 days if CrCL> 50 mL / min or 3 to 5 days if CrCL <50 mL / min before the procedure
* Patient under desmopressin acetate (DDAVP)
* Patient with HIV or Hepatitis C positive or Hepatitis B infection, defined by either a detection of the HBs antigen or the presence of anti HBc antibodies without HBs antibody detectable.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Success rate of establishment of the organoid culture | 15 days
  The success rate is defined by the rate of successful cell culture. A Cell culture is successful when organoids grow from dividing cells

SECONDARY OUTCOMES:
Drugs testing on organoid for cell viability | 20 days
  Viable cell count in different cells culture conditions using Cell titer Glo and viable cell count using typan blue
Cell Apoptosis Molecular and cellular mechanisms of drugs responses | 20 days
  Apoptosis biomarkers analysis in microscopy. Caspase 3 will be assess using microspcopy .
Cell proliferation Molecular and cellular on mechanisms of drugs responses | 20 days
  Proliferative biomarkers analysis in microscopy. Ki67 will be assess using microspcopy .

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: No